CLINICAL TRIAL: NCT01879371
Title: Relative Bioavailability of Ibuprofen From a Fixed Dose Combination (FDC) Tablet of Ibuprofen 400 mg and Caffeine 100 mg Compared to a Tablet of Ibuprofen 400 mg and a Tablet of Ibuprofen Lysinate 400 mg Following Oral Administration in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Three-period Crossover Study)
Brief Title: Relative Bioavailability of Ibuprofen From a Single Fixed Dose Combination Tablet of Ibuprofen and Caffeine Compared to Single Tablets of Ibuprofen and Ibuprofen Lysinate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1335.2; 2013-000990-66 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ibuprofen

ARMS (3):
- Ibuprofen (Brufen®) (Active Comparator): film-coated tablet
  Interventions: Drug: Ibuprofen (Brufen®)
- Ibuprofen (Nurofen Immedia®) (Active Comparator): film-coated tablet
  Interventions: Drug: Ibuprofen (Nurofen Immedia®)
- Ibuprofen+caffeine (Experimental): fixed-dose-combination (FDC)
  Interventions: Drug: Ibuprofen+caffeine FDC

INTERVENTIONS:
Drug: Ibuprofen+caffeine FDC — oral dose
  Arms: Ibuprofen+caffeine
Drug: Ibuprofen (Nurofen Immedia®) — oral dose
  Arms: Ibuprofen (Nurofen Immedia®)
Drug: Ibuprofen (Brufen®) — oral dose
  Arms: Ibuprofen (Brufen®)

SUMMARY:
To investigate the relative bioavailability of ibuprofen from a (FDC) film-coated tablet of ibuprofen and caffeine vs. a tablet of ibuprofen (Brufen®) and a tablet of ibuprofen lysinate (Nurofen Immedia®).

ELIGIBILITY:
Inclusion criteria:

* Healthy male and female subjects
* Age 18 to 50 years
* Body mass index (BMI) 18.5 to 29.9 kg/m2
* Subjects must be able to understand and comply with study requirements

Exclusion criteria:

- Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1335.2.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 healthy male and female subjects (at least a third of each sex) were recruited from the volunteers' pool of the Human Pharmacology centre of BI Pharma GmbH & Co. KG, Ingelheim, Germany.
Groups:
- Ibu + Caf / Ibu Acid / Ibu Lysinate: Participants first received Treatment T (400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet). After a washout phase of at least 6 days, they then received Treatment R1 (400mg Ibuprofen acid (Brufen®) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment R2 (400mg Ibuprofen lysinate (Nurofen® immedia) film-coated tablet). Every treatment is given oral as single dose of one tablet with 240 mL of water after an overnight fast of at least 10 h.
- Ibu + Caf / Ibu Lysinate / Ibu Acid: Participants first received Treatment T (400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet). After a washout phase of at least 6 days, they then received Treatment R2 (400mg Ibuprofen lysinate (Nurofen® immedia) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment R1 (400mg Ibuprofen acid (Brufen®) film-coated tablet). Every treatment is given oral as single dose of one tablet with 240 mL of water after an overnight fast of at least 10 h.
- Ibu Acid / Ibu Lysinate/ Ibu + Caf: Participants first received Treatment R1 (400mg Ibuprofen acid (Brufen®) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment R2 (400mg Ibuprofen lysinate (Nurofen® immedia) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment T (400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet). Every treatment is given oral as single dose of one tablet with 240 mL of water after an overnight fast of at least 10 h.
- Ibu Acid/ Ibu + Caf / Ibu Lysinate: Participants first received Treatment R1 (400mg Ibuprofen acid (Brufen®) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment T (400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet). After a washout phase of at least 6 days, they then received Treatment R2 (400mg Ibuprofen lysinate (Nurofen® immedia) film-coated tablet). Every treatment is given oral as single dose of one tablet with 240 mL of water after an overnight fast of at least 10 h.
- Ibu Lysinate/ Ibu + Caf / Ibu Acid: Participants first received Treatment R2 (400mg Ibuprofen lysinate (Nurofen® immedia) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment T (400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet). After a washout phase of at least 6 days, they then received Treatment R1 (400mg Ibuprofen acid (Brufen®) film-coated tablet). Every treatment is given oral as single dose of one tablet with 240 mL of water after an overnight fast of at least 10 h.
- Ibu Lysinate / Ibu Acid / Ibu + Caf: Participants first received Treatment R2 (400mg Ibuprofen lysinate (Nurofen® immedia) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment R1 (400mg Ibuprofen acid (Brufen®) film-coated tablet). After a washout phase of at least 6 days, they then received Treatment T (400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet). Every treatment is given oral as single dose of one tablet with 240 mL of water after an overnight fast of at least 10 h.
Period: Overall Study
Arm/Group | Ibu + Caf / Ibu Acid / Ibu Lysinate | Ibu + Caf / Ibu Lysinate / Ibu Acid | Ibu Acid / Ibu Lysinate/ Ibu + Caf | Ibu Acid/ Ibu + Caf / Ibu Lysinate | Ibu Lysinate/ Ibu + Caf / Ibu Acid | Ibu Lysinate / Ibu Acid / Ibu + Caf
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): included all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibu + Caf / Ibu Acid / Ibu Lysinate | Ibu + Caf / Ibu Lysinate / Ibu Acid | Ibu Acid / Ibu Lysinate/ Ibu + Caf | Ibu Acid/ Ibu + Caf / Ibu Lysinate | Ibu Lysinate/ Ibu + Caf / Ibu Acid | Ibu Lysinate / Ibu Acid / Ibu + Caf | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (7.6) | 36.3 (3.3) | 42.8 (4.5) | 40.2 (3.8) | 37.5 (9.2) | 38.3 (7.1) | 39.0 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 2 | 2 | 0 | 15
  Male | 2 | 2 | 3 | 4 | 4 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tz)
Description: AUC(0-tz): area under the concentration-time curve of Ibuprofen in plasma over the time interval from 0 to the last quantifiable data point
Time Frame: 2 hours (h) before drug administration and 5minutes (min), 10min, 15min, 30min, 45min, 1h, 1h 15min, 1h 30min, 1h 45min, 2h, 2h 30min, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h after drug administration
Population: Pharmacokinetic set (PKS): included all treated subjects who provided at least one observation for at least one primary Pharmacokinetic endpoint without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Groups:
- Ibuprofen + Caffeine (FDC) Tablet: 400 mg Ibuprofen + 100 mg Caffeine fixed dose combination (FDC) tablet; Single dose oral administration of one tablet with 240 mL of water after an overnight fast of at least 10h
- Ibuprofen Acid Film-coated Tablet: 400 mg Ibuprofen acid (Brufen®) film-coated tablet; Single dose oral administration of one tablet with 240 mL of water after an overnight fast of at least 10h
- Ibuprofen Lysinate Film-coated Tablet: Ibuprofen lysinate (Nurofen® immedia) film-coated tablet; 400 mg Ibuprofen; Single dose oral administration of one tablet with 240 mL of water after an overnight fast of at least 10h
Arm/Group | Ibuprofen + Caffeine (FDC) Tablet | Ibuprofen Acid Film-coated Tablet | Ibuprofen Lysinate Film-coated Tablet
Number analyzed (Participants) | 36 | 36 | 36
μg*h/mL | 133 (22.2) | 124 (19.4) | 122 (19.3)
Statistical Analysis 1: Comparison: Ibuprofen + Caffeine (FDC) Tablet vs Ibuprofen Acid Film-coated Tablet; The ANOVA (analysis of variance) model on the logarithmic scale included effects accounting for the following sources of variation: 'sequence', 'period' and 'treatment' as fixed effects and 'subjects within sequences' as random effect. The main focus was on estimation and not on testing, that is, formal statistical hypotheses were not tested; Test type: Superiority or Other; Geometric mean ratio (net) = 107.85, 90% CI 2-sided [105.334 to 110.431] — The geometric mean ratio is calculated as the geometric mean of 'Ibuprofen + Caffeine (FDC) tablet ' divided by the geometric mean of ' Ibuprofen acid film-coated tablet '
Statistical Analysis 2: Comparison: Ibuprofen + Caffeine (FDC) Tablet vs Ibuprofen Lysinate Film-coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio (net) = 109.48, 90% CI 2-sided [107.072 to 111.936] — The geometric mean ratio is calculated as the geometric mean of 'Ibuprofen + Caffeine (FDC) tablet ' divided by the geometric mean of ' Ibuprofen lysinate film-coated tablet '

2. Primary Outcome: Cmax
Description: Cmax: maximum measured concentration of Ibuprofen in plasma
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Ibuprofen + Caffeine (FDC) Tablet | Ibuprofen Acid Film-coated Tablet | Ibuprofen Lysinate Film-coated Tablet
Number analyzed (Participants) | 36 | 36 | 36
μg/mL | 31.0 (17.2) | 31.1 (22.5) | 44.0 (20.6)
Statistical Analysis 1: Comparison: Ibuprofen + Caffeine (FDC) Tablet vs Ibuprofen Acid Film-coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio (net) = 99.65, 90% CI 2-sided [93.874 to 105.776] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ibuprofen + Caffeine (FDC) Tablet vs Ibuprofen Lysinate Film-coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio (net) = 70.42, 90% CI 2-sided [67.087 to 73.928] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: AUC(0-inf)
Description: AUC(0-inf): area under the concentration-time curve of Ibuprofen in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Ibuprofen + Caffeine (FDC) Tablet | Ibuprofen Acid Film-coated Tablet | Ibuprofen Lysinate Film-coated Tablet
Number analyzed (Participants) | 35 | 36 | 36
μg*h/mL | 135 (21.7) | 127 (20.1) | 125 (20.2)
Statistical Analysis 1: Comparison: Ibuprofen + Caffeine (FDC) Tablet vs Ibuprofen Acid Film-coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio (net) = 106.50, 90% CI 2-sided [104.050 to 109.004] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Ibuprofen + Caffeine (FDC) Tablet vs Ibuprofen Lysinate Film-coated Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio (net) = 108.59, 90% CI 2-sided [106.185 to 111.054] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: from up to 21 days prior to first drug administration until 30 days after end of trial, 64 days
Arm/Group | Ibuprofen + Caffeine (FDC) Tablet | Ibuprofen Acid Film-coated Tablet | Ibuprofen Lysinate Film-coated Tablet
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 2/36 | 4/36 | 1/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen + Caffeine (FDC) Tablet (N=36) | Ibuprofen Acid Film-coated Tablet (N=36) | Ibuprofen Lysinate Film-coated Tablet (N=36)
Headache (Nervous system disorders) | 2 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes